CLINICAL TRIAL: NCT07372092
Title: Surgical Geriatrics o Geriatric Surgery? Outcomes in a Novel Hospital Model of Attention. A Comparative Cohort Study.
Brief Title: Complications of Surgical Geriatrics Hospitalized in the Orinoco Region
Acronym: SURGER
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital Departamental de Villavicencio (Other)
Collaborators: Cooperative University of Colombia (Other)
Responsible Party: Principal Investigator, Norton Perez-Gutierrez, MD, ICU director, Hospital Departamental de Villavicencio
Other Study IDs: GRIVI_2026_01_SURG_GERIATRICS
Record Dates: First submitted 2026-01-20; First posted 2026-01-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Operative Surgical Procedures; Aged; Aged 65 Years or Older; Geriatric; Geriatric Assessment; Postoperative Care; Postoperative Complications
Keywords: Operative Surgical Procedures; Aged; Geriatrics; Geriatric Assessment; Postoperative Care; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- First period: Period previous to the implementation of the geriatric surgical program
  Interventions: Other: Hip fractures
- Second period: Period posterior to the implementation of a geriatric surgical program

INTERVENTIONS:
Other: Hip fractures — Geriatric patients with surgical operations for hip fractures or colonic diverticular disease previos or posterior to the implementation of a geriatric surgical program
  Groups: First period

SUMMARY:
The life expectancy of the Colombian population is increasing. Older patients are frequently hospitalized and treated in surgical wards, and are treated as the general surgical population. However, geriatric patients are frequently found with additional comorbidities, besides the primary surgical diagnosis. Some diseases, like hip fractures, diverticulitis, and cancer, are common in this age range. The preoperative, intraoperative, and postoperative period requires a special care and planning to avoid complications related to the physical status, medications, and comorbidities. Studies about the geriatric surgical population are limited in the Orinoco region. The implementation of a comprehensive geriatric assesment in surgical services requires follow-up of outcomes.

DETAILED DESCRIPTION:
Introduction: The increase in patients' life expectancy increases the likelihood that older adults will undergo surgical procedures. This underscores the need for comprehensive care that considers the special needs of this age group, delivered by a collaborative team, to achieve improved outcomes and provide quality care. The aim of the study is to compare the factors associated with adverse outcomes in geriatric patients undergoing surgical procedures.

Methodology: An observational, retrospective cohort study will be conducted at the Hospital Departamental de Villavicencio and the Clinica Primavera between August 2026 and July 2027. Discharged records of older adult patients (65 years and older) admitted to surgical specialties, both emergency and elective, will be included. Patients with the codes S720, S324, S730, S731, S770, S772, S797, and S798 in the tenth edition of the International Classification of Diseases (ICD 10th) will be included. Patients with the codes K472, K573, K574, K758, and K579 will also be included. These codes were slected as hip fractures and colonic diverticular disease are typical in older adults. The outcomes to be studied will be mortality, length of hospital stay, need for ICU admissions, and ICU length of stay. Study variables will include demographic data, surgical diagnosis, surgical specialty, comorbidities, and complications, as defined by the Clavien-Dindo classification. A comparison of the cohort before and after the implementation of a surgical and geriatric program will be performed.

ELIGIBILITY:
Inclusion Criteria:

* Adults
* Hospitalized in the surgical ward
* Surgical procedures

Exclusion Criteria:

* Derived to other institution
* Operated previously in other institution

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adults discharged from the surgical wards in the study period.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2027-07-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 28 days
  All-cause mortality within 28 days of the surgical procedure

SECONDARY OUTCOMES:
Complications | 28 days
  Complications within 28-days of the surgical procedure

CONTACTS AND LOCATIONS:
Overall Officials: Norton Perez, Principal Investigator — Hospital Departamental de Villavicencio
Locations (1):
- Hospital Departamental de Villavicencio, Villavicencio, Meta Department, Colombia

IPD SHARING:
Plan to Share IPD: Undecided
It contains sensitive information about patients.

REFERENCES:
- [Background] Pugliese M, Connell L, Turco J, Trivedi A, Foster A, Kumarasinghe APW. Implementation of a geriatric in-reach service improves acute surgical unit outcomes; a retrospective before-and-after study. ANZ J Surg. 2024 Jul-Aug;94(7-8):1349-1355. doi: 10.1111/ans.19026. Epub 2024 May 10. PMID 38727023
- [Background] Sagona A, Ortega CA, Wang L, Brameier DT, Selzer F, Zhou L, von Keudell A. Frailty Is More Predictive of Mortality than Age in Patients With Hip Fractures. J Orthop Trauma. 2024 Aug 1;38(8):e278-e287. doi: 10.1097/BOT.0000000000002844. PMID 39007664
- [Background] Ding L, Tao X, Zhou J. Effect of a comprehensive geriatric assessment-based individualized intervention on postoperative patients with cerebral hemorrhage: A randomized controlled study. Technol Health Care. 2024;32(3):1555-1567. doi: 10.3233/THC-230611. PMID 38073343
- [Background] Jones TS, Peters X, Robinson TN. Clin-STAR corner: Practice-changing advances at the interface of surgery and geriatrics. J Am Geriatr Soc. 2024 Jul;72(7):1959-1963. doi: 10.1111/jgs.18783. Epub 2024 Jan 27. PMID 38280226
- [Background] Boukebous B, Biau D, Gao F. AtoG: A simple score to predict complications and death after hip fractures, in line with the comprehensive geriatric assessment. Orthop Traumatol Surg Res. 2024 May;110(3):103827. doi: 10.1016/j.otsr.2024.103827. Epub 2024 Jan 26. PMID 38280714
- [Background] Arcidiacono GP, Ceolin C, Sella S, Camozzi V, Bertocco A, Torres MO, Roda MG, Cannito M, Berizzi A, Romanato G, Venturin A, Cianci V, Pizziol A, Pala E, Cerchiaro M, Savino S, Tessarin M, Simioni P, Sergi G, Ruggieri P, Giannini S; Hip-POS working group. Taking care of inpatients with fragility hip fractures: the hip-padua osteosarcopenia (Hip-POS) fracture liaison service model. J Endocrinol Invest. 2025 Jan;48(1):99-108. doi: 10.1007/s40618-024-02425-z. Epub 2024 Jul 6. PMID 38971949
- [Background] Choi JY, Park JW, Kim KI, Lee YK, Kim CH. Prediction of 5-Year Survival Rate After Hip Fracture Surgery Using a Comprehensive Geriatric Assessment-Based Frailty Score Model. J Korean Med Sci. 2025 Mar 31;40(12):e40. doi: 10.3346/jkms.2025.40.e40. PMID 40165573
- [Background] Jimenez-Mola S, Plaza-Carmona M, Idoate Gil FJ, Saez-Lopez P, Fernandez Garcia P, Seco-Calvo J. Functional decline in nonagenarians admitted for hip fracture. Rev Assoc Med Bras (1992). 2025 Mar 17;71(1):e20240796. doi: 10.1590/1806-9282.20240796. eCollection 2025. PMID 40105545